CLINICAL TRIAL: NCT06291740
Title: Continuous Versus Intermittent Nebulization Therapy in Acute Asthma Exacerbation at Emergency Department: A Randomized Controlled Trial
Brief Title: Continuous Versus Intermittent Nebulization Therapy in Acute Asthma Exacerbation at Emergency Department
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Kumpol Kornthatchapong, Associated Professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-EM-2-008/67; Faculty of Medicine (Other: Thammasat University, Thailand)
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Asthma Exacerbation; Emergency Department; Nebulization
Keywords: asthma exacerbation; continuous nebulization; intermittent nebulization
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous nebulization (Experimental): continuous nebulization using the MiniHEART-HiFlo® nebulizer containing Budesonide 1000 microgram/2 ml (3 respules) + 1.25 mg of fenoterol and 0.5 mg of ipratropium bromide (Berodual®, 4 ml) and Normal saline 12 ml in the nebulizer chamber. Patients in this group will receive continuous aerosol therapy over a period of 1 hour at an oxygen flow rate of 8 L/min
  Interventions: Device: continuous nebulization
- intermittent nebulization (Active Comparator): intermittent nebulization using a nebulizer containing Budesonide 1000 microgram/2 ml (1 respules) + 1.25 mg of fenoterol and 0.5 mg of ipratropium bromide (Berodual®, 4 ml) at an oxygen flow rate of 10 L/min every 20 minutes, thrice within 1 hour
  Interventions: Device: Intermittent nebulization

INTERVENTIONS:
Device: continuous nebulization — continuous nebulization using the MiniHEART-HiFlo® nebulizer containing Budesonide 1000 microgram/2 ml (3 respules) + 1.25 mg of fenoterol and 0.5 mg of ipratropium bromide (Berodual®, 4 ml) and Normal saline 12 ml in the nebulizer chamber. Patients in this group will receive continuous aerosol therapy over a period of 1 hour at an oxygen flow rate of 8 L/min
  Arms: Continuous nebulization
Device: Intermittent nebulization — intermittent nebulization using a nebulizer containing Budesonide 1000 microgram/2 ml (1 respules) + 1.25 mg of fenoterol and 0.5 mg of ipratropium bromide (Berodual®, 4 ml) at an oxygen flow rate of 10 L/min every 20 minutes, thrice within 1 hour
  Arms: intermittent nebulization

SUMMARY:
The goal of this clinical is to compare treatment outcomes between continuous nebulization and intermittent therapy in the management of acute exacerbation of asthma in the emergency department(ED). Participants will random assign to either continuous or intermittent nebulization. In the continuous group, patients receive budesonide, fenoterol, ipratropium bromide, and normal saline continuously for an hour. In the intermittent group, the same medications are administer every 20 minutes for an hour. Measurements include symptom severity, respiratory rate, oxygen saturation, and pulmonary function tests. Primary endpoints are ED stay length, hospital admission, and ED revisit within 48 hours post-discharge. Adverse events are documented.

ELIGIBILITY:
Inclusion Criteria:

* asthma exacerbation

Exclusion Criteria:

* life-threatening conditions requiring intubation
* allergy to steroid or its components
* patient under investigation of Corona Virus Disease, 2019 (COVID-19)
* pulmonary tuberculosis
* unable to cooperate for pulmonary function testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Length of ED stay | through study completion, an average of 1 year
  duration of ED management

SECONDARY OUTCOMES:
pulmonary function test | through study completion, an average of 1 year
  Forced Expiratory Volume in one second(FEV1), Peak Expiratory Flow(PEF)

OTHER OUTCOMES:
Hospital admission | through study completion, an average of 1 year
ED revisit within 48 hours | through study completion, an average of 1 year
  revisit with acute asthma exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Kumpol Kornthatchapong, Principal Investigator — Faculty of Medicine, Thammasat university

REFERENCES:
- See also: Comparison of intermittent and continuously nebulized albuterol for treatment of asthma in an urban emergency department — https://pubmed.ncbi.nlm.nih.gov/8239105/
- See also: Continuous versus intermittent albuterol nebulization in the treatment of acute asthma — https://pubmed.ncbi.nlm.nih.gov/8239106/
- See also: A randomized, clinical trial comparing the efficacy of continuous nebulized albuterol (15 mg) versus continuous nebulized albuterol (15 mg) plus ipratropium bromide (2 mg) for the treatment of acute asthma — https://pubmed.ncbi.nlm.nih.gov/17046476/